CLINICAL TRIAL: NCT04162977
Title: Well-Venture Pilot Project: Adapting Personality-Targeted Interventions for Reducing Substance Misuse and Related Outcomes in Youth in Youth Protection Services
Brief Title: Adapting Personality-Targeted Interventions for Reducing Substance Misuse and Related Outcomes in Youth in Youth Protection Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Batshaw Youth and Family Centres (Unknown)
Responsible Party: Principal Investigator, Hanie Edalati, Postdoctoral Fellow, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Well-Venture Project
Record Dates: First submitted 2019-08-19; First posted 2019-11-14 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Substance Use Disorders; Youth Protection Services; Early Intervention; Prevention; Adolescent Development
Keywords: Substance Use and Misuse; Prevention; Early Intervention; Mental Health; Complex Trauma; Youth Protection Services.; Adolescence; Personality-targeted Interventions
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study examines the feasibility and proof-of-concept of implementing personality-targeted interventions for high-risk adolescents receiving services from Youth Protection Services. For testing the feasibility, this study compares the following outcomes with the same outcomes from previous Preventure trials with community samples: facilitator's score on Intervention/implementation fidelity, number of high-risk youth who agree to participate in intervention sessions, and elements of youth's feedback. For testing the proof-of-concept, this study examines effects of interventions on change in substance use outcomes, depression symptoms, and self-reported anxiety sensitivity and impulsivity at 3- and 6-month post-intervention. Previous trials with the community samples indicated that these primary outcomes largely accounted for the long-term intervention effects on reduction of substance use outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-risk youth (Experimental): The 23-item Substance Use Risk Profile Scale (SURPS) will be used to identify high-risk adolescents who enter the intervention trial. Adolescents who score high on one of SURPS subscales (i.e., high-risk youth) will be invited to participate in two group-based intervention sessions which target their dominant personality profile. The criterion for high scores on SURPS personality traits are determined based on norms from high-risk adolescents in the same age range who participated in previous trials on personality-targeted interventions.
  Interventions: Behavioral: Personality-targeted Interventions

INTERVENTIONS:
Behavioral: Personality-targeted Interventions — The Personality-targeted Interventions (i.e., Preventure programme) are selective substance use prevention programme designed to target known personality risk factors for substance misuse based on the evidence from cross-sectional and longitudinal studies which connect these personality risk factors to early initiation and escalation of substance misuse in adolescents. This selected personality-targeted approach targets four personality-specific motivational pathways to substance misuse: Hopelessness, Anxiety Sensitivity, Impulsivity, and Sensation Seeking. Each intervention will involve two 90-minute sessions, with an average of 6 personality-matched adolescents per group, and will be conducted using manuals that incorporate psycho-educational, motivational enhancement therapy (MET), and cognitive behavioural therapy (CBT) components and include real life 'scenarios' shared by high-risk local youth with similar personality profiles.
  Other Names: Preventure programme

SUMMARY:
Substance use problems are major concern in adolescents involved in Youth Protection Services. However, there is an enormous gap between the needs and availability of interventions for youth with substance use problems in the system. The present study will examine the feasibility and proof-of-concept of implementing an evidence-based, personality-targeted drug and alcohol prevention programme for high-risk adolescents (i.e., Preventure programme) receiving services from Youth Protection Services. Our goal is to examine the effects of these interventions on reducing rates of substance use outcomes, depression symptoms, and self-reported anxiety sensitivity and impulsivity at 3- and 6-month post-intervention. These primary outcomes were selected based on previous Preventure trials with the community samples, that indicated these factors largely accounted for the long-term intervention effects on improving substance use outcomes. The study will be conducted at Batshaw Youth and Family Centres, which provide psychosocial, rehabilitation and social integration services and services related to child placement and adoption to English-speaking youth from all regions of Quebec. Adolescents receiving services from Batshaw centres (N = 100, aged 14 and above) will be invited to participate in the study. All interested adolescents will be invited to attend one assessment session with the research team. Participants who score high on one of subscales of Substance Use Risk Profile Scale (SURPS) (i.e., high-risk adolescents) will be invited to participate in two 90-minute group-based intervention sessions, which target their dominant personality profile. Sessions will be cognitive-behavioural in nature and are designed to help youth understand the target personality trait and develop adaptive coping strategies for managing that trait using motivational and cognitive restructuring techniques. The primary outcomes will be measured at baseline before receiving the interventions and then with 3-month and 6-month intervals after receiving the interventions to test whether these outcomes are significantly reduced after receiving the interventions. The results of this study will be used to plan the future directions of personality-targeted interventions for youth involved in Youth Protection Services.

DETAILED DESCRIPTION:
Background and aims

Substance use problems are major concern in adolescents involved in Youth Protection Services. Some studies estimated that 1 in 5 adolescents involved in Youth Protection Services struggle with a substance use problem. In addition, living in foster homes increases the likelihood of substance abuse by five times compared to no history of removal. Investigators of this study have conducted a review to identify the gaps in research and service delivery for substance use prevention and early interventions among at-risk adolescents involved in Youth Protection Services. This review showed that there is an enormous gap between the needs and availability of interventions for youth with substance use problems with less than 10% of these adolescents and young adults receive such interventions. This article also reviewed the evidence that showed targeting personality risk profiles is potentially a good strategy for reducing substance use problems and increasing resilience in this population.

The present study examines the feasibility and proof-of-concept of implementing an evidence-based, personality-targeted drug and alcohol prevention programme (i.e., Preventure programme) for high-risk adolescents receiving services from Youth Protection Services.The Preventure programme is a selective substance use prevention programme designed to target known personality risk factors for substance misuse based on the evidence from cross-sectional and longitudinal studies which connect these personality risk factors to early initiation and escalation of substance misuse in adolescents. This selected personality-targeted approach targets four personality-specific motivational pathways to substance misuse: Hopelessness (Negative Thinking), Anxiety Sensitivity, Impulsivity and Sensation Seeking.

The study is conducted at Batshaw Youth and Family Centres, which provide psychosocial, rehabilitation and social integration services and services related to child placement and adoption to English-speaking youth from all regions of Quebec.

A working group consisting of research scientists in the fields of adolescent mental health, childhood trauma, and substance use prevention and the coordinator of the residential and rehabilitation program of Batshaw Centres, met on February 11, 2019 to discuss details of the pilot trial, required changes to the content of personality-targeted interventions (i.e., Preventure Programme), and the study timeline.

Study Design

Participants. All adolescents receiving services from the Batshaw Centres, starting October 2nd, 2019, are invited to participate in this study. Batshaw Centres provide services to an average of 100 adolescents aged 14 and above during every 6-month period. This study aims to recruit all interested adolescents aged 14 and above for this pilot project.

Recruitment & Consent. Staff at Batshaw Centres will give a brief description including basic information about the study to all adolescents in their units. Interested participants will be invited for the pre-intervention screening. Passive consent from parents or legal guardians is required. Prior to starting the study, an information letter will be provided to all parents notifying them that the study is taking place at Batshaw Centres and explaining the study and interventions. They will be asked to sign and return the letter if they do not agree to their child participating in this study. An assent form will be provided to adolescents and thoroughly explained by the Batshaw staff and research investigator. Adolescents are required to sign the assent form prior starting the study.

Procedure. Adolescents who score high on one of the Substance Use Risk Profile Scale (SURPS) (i.e., high-risk individuals) will be invited to participate in brief group-based intervention sessions which target their dominant personality profile. The criterion for high scores on SURPS personality traits (i.e., high-risk) are determined based on norms from high-risk adolescents in the same age range who participated in previous trials of personality-targeted interventions. Intervention sessions will be delivered by trained educators or counsellors from Batshaw. According to the literature, it is estimated that around 80% of recruited youth (N ~ 80) will show high scores in one of the personality risk profiles. The rest of participants (N ~ 20; low-risk adolescents) will receive the treatment as usual. Adolescents receive an honorarium of $30 in the form of gift card upon completion of each assessments for a total of $90.

Screening. Both groups of participants will be followed for 6 months. Screening will take place using a computerized program installed on laptops provided by the research team. The screening is completed at baseline and then 3-month and 6-month intervals after receiving the interventions and takes 50-60 minutes. The screening procedure includes several questionnaires and computerized tasks, which have been validated by the scientific community. These questionnaires involve assessing youth's personality traits, cognitive functioning, substance use outcomes, and psychiatric symptoms. The research investigator will be present during the assessment sessions to ready the participants and materials, give instructions, expla study goals and procedure, answer questions and supervise the session.

Outcome Measures. All participants will be assessed by the same measures 3 and 6 months after receiving the interventions.

For testing the feasibility, this study will compare the following outcomes with the same outcomes from the previous successful trials with the community samples: facilitator's score on Intervention/implementation fidelity, number of high-risk youth who agree to participate in the intervention sessions, and elements of youth's feedback (assessment immediately at the end of second intervention session). Preventure Intervention/implementation Fidelity Scale (PIFA) was designed by the Preventure team to measure the level of implementation of the programme and facilitators' adherence and fidelity to the critical ingredients of the Preventure programme. This measure has been used in previous trials of Preventure programme with the community samples. Group Experience Questionnaire was also designed by the Preventure team to measure youth-generated perspectives and feedback on the intervention. Our previous studies using this questionnaire have shown that youth perspectives on the intervention independently accounted for up to 12-25% of the variance in changes in alcohol consumption and mental health symptoms over 12 months. These findings highlight the positive youth experiences of the programme as a significant indicator of its efficacy.

For the proof-of-concept, this study will examine the rates of depression symptoms, self-reported anxiety sensitivity and impulsivity and several substance use outcomes at baseline and then 3-month and 6-month intervals after receiving the interventions and test whether these outcomes are significantly reduced after receiving the interventions. These primary outcomes (i.e., early mechanisms of change) were selected based on previous Preventure trials with the community samples, that indicated these factors largely accounted for the long-term intervention effects on improving substance use outcomes. According to our conversation with the Batshaw centres, around 60% of the adolescents in their care suffer from some forms of substance use problems. Therefore, reductions in substance use problems is regarded as a significant indicator of the proof-of-concept in this study.

Additional information on research participants. The rates of childhood adversity/maltreatment, involvement in criminal justice system, low academic performance, and psychiatric diagnoses are particularly high in this population, which may influence the results of the study. In addition, the exact date of the admission and type of other interventions received before and during this trial are needed to be considered in the analyses. Participants' files will be used to gain this information. A protocol was designed, and approved by the Research Ethics Board to access participants' files.

Interventions. All interventions will be conducted at Batshaw centres by a trained facilitator and a co-facilitator. After selection on personality scale (i.e., SURPS), high-risk adolescents will be invited to participate in brief group-based intervention sessions which target their dominant personality profile (Hopelessness, Anxiety Sensitivity, Impulsivity, or Sensation Seeking). Each intervention will involve two 90-minute sessions, with an average of 4-6 personality-matched adolescents per group, and will be conducted using manuals that incorporate psycho-educational, motivational enhancement therapy (MET), and cognitive behavioural therapy (CBT) components which include real life 'scenarios' shared by high-risk youth from Montreal with similar personality profiles.

Analyses. Correlation analyses will be used to examine the patterns of substance use and related mental health problem in relation to personality profiles of adolescents in Youth Protection Services. For the feasibility analyses, t-test will be used to compare results of facilitator's score on Intervention/implementation fidelity scale, number of high-risk youth who agree to participate in the interventions, and elements of youth's feedback with results from previous trials which were successful in reducing rates of substance use outcomes among community samples. For proof-of-concept analyses, a repeated measure ANCOVA will be used to examine the change in pre- and post-intervention assessments of substance use outcomes, depression symptoms, and scores of anxiety sensitivity and impulsivity while controlling for the effects of confounding variables such as histories of childhood maltreatment and socio-economic status. This study will also conduct some secondary data analyses with other outcomes such as cognitive functioning, and psychiatric symptoms to guide future directions.

Follow-up survey. After completing the intervention sessions, some of youth who received personality-targeted interventions and group facilitators will be invited to participate in separate focus groups with the research team to comment on various aspects of their experiences of interventions using a qualitative method. This qualitative data and the quantitative data from the pre- and post-intervention assessments will be discussed in the second working group to plan the future directions for personality-targeted interventions for youth involved in Youth Protection Services.

ELIGIBILITY:
Inclusion Criteria:

• Receiving services from Batshaw Youth and Family Centres under the Youth Protection Services

Exclusion Criteria:

* Severe cognitive impairments
* Acute psychotic symptoms

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Rate of Depression Symptoms | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of depression symptoms is assessed using depression subscale of Brief Symptom Inventory. The depression subscale includes six items each rated on a five-point scale (0 = not at all, 1 = a little bit, 2 = moderately, 3 = quite a bit, 4 = often). Responses are summed to create a total score ranging from 0 to 24. Higher scores indicate higher rates of depression symptoms.
Self-reported Anxiety Sensitivity | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the score of personality trait of anxiety sensitivity is assessed using anxiety sensitivity subscale of Substance Use Risk Profile Scale. Substance Use Risk Profile Scale assesses the variability on the four personality risk factors for substance misuse and dependence. Anxiety sensitivity subscale includes 5 items rated on a 4 point scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Responses are summed to create a total score ranging from 5 to 20. Higher scores indicate more elevation on personality trait of anxiety sensitivity.
Feasibility Outcome 1: Score on Preventure Intervention/implementation Fidelity Scale | Baseline during two intervention sessions
  Facilitator's score on Preventure Intervention/implementation Fidelity Scale (PIFA) rated by session supervisor: Preventure Intervention/implementation Fidelity Scale (PIFA) evaluates adherence to 12 core treatment components of the personality-targeted intervention program (e.g., goal setting, identifying and challenging automatic thoughts). This scale will be used during supervision in order to provide trainees with feedback and ensure that they reached sufficient levels of program delivery.
Feasibility Outcome 2: Number of high-risk youth who agree to participate in the intervention sessions | Baseline
  Number of high-risk youths who agree to participate in the intervention sessions.
Feasibility Outcome 3: Youth-generated feedback | Baseline (directly post-intervention)
  Percentage of youth reporting positive group experiences, learning and skill development: Participants will complete a brief feedback questionnaire regarding their intervention experiences directly following the final intervention session. This questionnaire includes 22 questions asking about their experiences of participating in the workshops rated on a 4-point scale ranging from Strongly Disagree to Strongly Agree. Participants will also respond to 4 open-ended questions in free format namely "Something that you liked about the group", "Something that you didn't like the group", "What is the most important thing you have learned from this workshop?" and "What is the change that you are considering?" Finally they will respond to questions relating to their level of motivation and self-efficacy to make a personal change using a 7-point Likert scale (0 = not at all motivated/confident, 7 = extremely motivated/confident).
Rate of Binge Drinking | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of binge drinking is assessed by an item from the 'Detection of alcohol and drug problems in adolescents' questionnaire (DEP-ADO). Binge drinking is assessed by asking youth to indicate how often they consumed five or more standard alcoholic drinks on the same occasion during the last 12 months (at baseline) or 3 months (at 3- and 6-month post-intervention assessments). Higher numbers indicate higher rate of binge drinking.
Total Number of Drug Used | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the total number of drug used is assessed by items from the 'Detection of alcohol and drug problems in adolescents' questionnaire (DEP-ADO). Youth are first asked to indicate if they have used one or more of the listed substances (e.g., Cannabis, Cocaine, Heroin, Opiates) and if so, to indicate how often they had consumed each in the past 12 months (at baseline) or 3 months (at 3- and 6-month post-intervention assessments) on a six-point scale (0 = never to 5 = every day). Higher scores indicate higher number of drug used.
Rate of Alcohol-related Harm | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of alcohol-related harm is assessed by items from the 'Detection of alcohol and drug problems in adolescents' questionnaire (DEP-ADO). As participants are encouraged to discuss their substance use problem as part of the intervention, the item from the original measure asked 'if they discussed their alcohol use with a counsellor in the last 12 months' will be removed from the analysis. Youth are asked to indicate if they have experienced any of the 9 listed problematic situations because of alcohol in the past 12 months (at baseline) or 3 months (at 3- and 6-month post-intervention assessments). Responses are rated as 1 = Yes and 0 = No and summed to create a total score ranging from 0 to 9. Higher scores indicate higher rates of alcohol-related harm.
Self-reported Impulsivity | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the score of personality trait of impulsivity is assessed using impulsivity subscale of Substance Use Risk Profile Scale. Substance Use Risk Profile Scale assesses the variability on the four personality risk factors for substance misuse and dependence. Impulsivity subscale includes 5 items rated on a 4 point scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Responses are summed to create a total score ranging from 5 to 20. Higher scores indicate more elevation on personality trait of impulsivity.
Rate of Drug-related Harm | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of drug-related harm is assessed by items from the modified version of 'Detection of alcohol and drug problems in adolescents' questionnaire (DEP-ADO). As participants are encouraged to discuss their substance use problem as part of the intervention, the item from the original measure asked 'if they discussed their drug use with a counsellor in the last 12 months' will be removed from the analysis. Youth are asked to indicate if they have experienced any of the 9 listed problematic situations because of drugs in the past 12 months (at baseline) or 3 months (at 3- and 6-month post-intervention assessments). Responses are rated as 1 = Yes and 0 = No and summed to create a total score ranging from 0 to 9. Higher scores indicate higher rates of drug-related harm.

SECONDARY OUTCOMES:
Rate of Anxiety Symptoms | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of anxiety symptoms is assessed using anxiety subscale of Brief Symptom Inventory. The anxiety subscale includes six items each rated on a five-point scale (0 = not at all, 1 = a little bit, 2 = moderately, 3 = quite a bit, 4 = often). Responses are summed to create a total score ranging from 0 to 24. Higher scores indicate higher rates of anxiety symptoms.
Emotion Dysregulation | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the total and dimensions scores of emotion dysregulation is measured by the Difficulties in Emotion Regulation Scale-Short Form (DERS-18). This scale consists of 18-items rated on a 5-point scale, from 1 (almost never) to 5 (almost always). Items capture six dimensions of emotion dysregulation: non-acceptance of emotional responses, difficulties engaging in goal-directed behaviour, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Responses are summed to create a total score of emotion dysregulation ranging from 18 to 90. Three items for each dimension subscale are summed to create a total score for that dimension ranging from 3 to 15. Higher scores indicate higher more emotion dysregulation problems.
Self-esteem Score | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the score of self-esteem is assessed using Rosenberg Self-Esteem Scale. Rosenberg Self-Esteem Scale assesses global self-worth by measuring both positive and negative feelings about the self. The scale consists of 10 items rated on a 4-point Likert scale ranging from 0=strongly disagree to 3=strongly agree. Responses are summed to create a total score ranging from 0 to 30. Higher scores indicate higher self-esteem.
Rate of Conduct Problems | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of conduct symptoms is assessed using conduct problem subscale of Strengths and Difficulties Questionnaire. The conduct problem subscale includes five items each rated on a three-point scale (0 = not true, 1 = sometimes true, 2 = certainly true). Responses are summed to create a total score ranging from 0 to 10. Higher values represent higher rates of conduct symptoms.
Rate of Hyperactivity/inattentive Problems | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of hyperactivity/inattentive symptoms is assessed using hyperactivity/inattentive subscale of Strengths and Difficulties Questionnaire. The hyperactivity/inattentive includes five items each rated on a three-point scale (0 = not true, 1 = sometimes true, 2 = certainly true). Responses are summed to create a total score ranging from 0 to 10. Higher values represent higher rates of hyperactivity/inattentive symptoms.
Rate of Post-traumatic Stress Disorder Symptoms | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of post-traumatic stress disorder (PTSD) symptoms is measured using the International Trauma Questionnaire for the International Classification of Diseases 11th Revision (ICD-11). Participants are first asked to identify 'the experience that troubles them most' and briefly describe it and then to respond to 9 items asking about their problems (i.e. symptoms) in the past month related to the experience. Responses are rated on a five-point scale (0 = not at all to 5 = extremely). A diagnosis of PTSD requires the endorsement of one of two symptoms from the symptom clusters of (1) reexperiencing in the here and now, (2) avoidance, and (3) sense of current threat, plus endorsement of at least one indicator of functional impairment associated with these symptoms. Endorsement of a symptom or functional impairment item is defined as a score of ≥ 2.
Rate of Complex-Post-traumatic Stress Disorder Symptoms | Baseline (pre-intervention), 3-month post-intervention, and 6-month post-intervention
  Change in the rate of complex-post-traumatic stress disorder (CPTSD) symptoms is measured using the International Trauma Questionnaire for the International Classification of Diseases 11th Revision. Participants are first asked to identify and briefly describe 'the experience that troubles them most' and then to respond to 18 items asking about their symptoms in the past month related to the experience on a five-point scale (0 = not at all to 5 = extremely). These items evaluate PTSD symptoms and disturbances in self-organization symptoms. A diagnosis of CPTSD requires the endorsement of one of two symptoms of the three PTSD symptoms clusters and one of two symptoms of the three disturbances in self-organization clusters. Endorsement of at least one indicator of functional impairment related to PTSD symptoms and one related to the disturbances in self-organization symptoms is required. Endorsement of a symptom or functional impairment item is defined as a score ≥ 2.

CONTACTS AND LOCATIONS:
Overall Officials: Hanie Edalati, PhD, Principal Investigator — St-Justine Hospital, University of Montreal; Patricia J Conrod, PhD, Principal Investigator — St-Justine Hospital, University of Montreal
Locations (1):
- Batshaw Youth and Family Centres, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edalati H, Conrod PJ. A Review of Personality-Targeted Interventions for Prevention of Substance Misuse and Related Harm in Community Samples of Adolescents. Front Psychiatry. 2019 Jan 22;9:770. doi: 10.3389/fpsyt.2018.00770. eCollection 2018. PMID 30723431
- [Background] Edalati H, Conrod PJ. A review to identify gaps in research and service delivery for substance use prevention among at-risk adolescents involved in child welfare system: the promises of targeted interventions. International Journal of Child and Adolescent Resilience (2017) 5:20-39.
- [Background] Woicik PA, Stewart SH, Pihl RO, Conrod PJ. The Substance Use Risk Profile Scale: a scale measuring traits linked to reinforcement-specific substance use profiles. Addict Behav. 2009 Dec;34(12):1042-55. doi: 10.1016/j.addbeh.2009.07.001. Epub 2009 Jul 8. PMID 19683400
- [Background] Conrod PJ. Personality-Targeted Interventions for Substance Use and Misuse. Curr Addict Rep. 2016;3(4):426-436. doi: 10.1007/s40429-016-0127-6. Epub 2016 Nov 4. PMID 27909645